CLINICAL TRIAL: NCT07044284
Title: A Pilot Study Looking at the Use of Virtual Reality Mindfulness Fractals in Addressing Menopause Symptoms, Sexual Function, Cognitive Mindfulness and Well-being
Brief Title: The Effects of Fractal Mindfulness Virtual Reality on Menopause Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Metropolitan University (Other)
Responsible Party: Principal Investigator, Samantha Banbury, Principal Investigator, London Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ALondonUni
Record Dates: First submitted 2025-06-26; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Menopause
Keywords: fractal mindfulness; wellbeing; Cognitive mindfulness; Sexual functioning

STUDY DESIGN:
Intervention Model Description: An active and a delayed group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): Fractal Mindfulness Virtual Reality
  Interventions: Device: Fractal mindfulness recombination
- Delayed group (Active Comparator): Fractal Mindfulness Virtual Reality
  Interventions: Device: Fractal mindfulness recombination

INTERVENTIONS:
Device: Fractal mindfulness recombination — Immersive virtual reality using fractal mindfulness software

SUMMARY:
The study aimed to establish the effectiveness of an immersive mindfulness virtual reality intervention using fractal software for women experiencing menopausal symptoms.

It was hypothesised that post immersive virtual reality fractal mindfulness intervention would result in higher levels of sexual function, wellbeing and cognitive mindfulness with lower levels of menopause symptoms. It was further hypothesised that in physiological responses, the pulse rate would be lower post intervention per session and an overall reduction in pulse rate post intervention. An electroencephalogram will be used to monitor alpha and beta ratios.

DETAILED DESCRIPTION:
Menopause is both a biological and psychological milestone that signifies the end of a woman's reproductive capacity and typically occurs between the ages of 45 and 55. A multitude of physiological, emotional, cognitive, and sexual symptoms often accompany this transition.

Putting aside the standard biopsychosocial interventions to one side, an alternative approach gaining momentum, associated with supporting meditation and mindfulness practices, is the use of fractals. Fractals exhibit varying levels of repetition with a rate of pattern shrinkage between repetitions, denoted by the D value where research has shown that fractals can reduce stress levels by increasing alpha brain wave in the frontal area of the brain. Fractal mindfulness utilises self-similar, repetitive patterns found in fractals to promote relaxation and offers insights into our perception of reality. With fractal mindfulness, the focus is on the present moment. This idea has been linked to spirituality because it explains humans' universal and innate subconscious understanding of the world. Increased levels of meditation are often associated with higher alpha and theta brain oscillations. Furthermore, sound can support the meditative state through beat frequencies, which can be observed through physiological measures such as changes in heart rate, increased relaxation, and a hypnotic state. Therefore, when fractals and music are combined, they may arguably create a more powerful response that fosters meditative awareness.

Artificial fractals may include computer-generated fractals, which are becoming increasingly widespread due to the increased use of digital technology, as recursive algorithms are used to generate them. However, living conditions do not always permit a complete connection with fractals in nature, and perhaps the increasing use of technology and virtual reality could serve as a helpful alternative. Fractals have become more accessible and scalable through digital platforms, enabling their integration into mainstream healthcare.

Despite the growing interest in fractals and digital health, few studies have explored the intersection of these two areas with menopause. Based on the literature review, this exploratory study examined the impact of a novel, immersive fractal mindfulness intervention on menopause-related symptoms, as well as sexual function, cognitive mindfulness, and overall well-being. This study employed a mixed methods approach, evaluating symptom change both quantitatively through standardised questionnaires and qualitatively through open-ended survey responses. Heart rate and an electroencephalogram further placed the outcomes into context, particularly when examining alpha and beta ratios.

All participants received the same intervention and were assessed at three time points: baseline week 0, post intervention week 4, and follow up week 8 in a waitlist randomised controlled study, which included active and delayed groups consisting of nine participants in each group. This ensured that every participant received the intervention. Feedback was solicited through five open ended questions to gauge the participants' perceptions of their experiences with the intervention. Pulse rate was recorded both before and after the session, and a basic electroencephalogram was employed to determine any increase in alpha waves in the occipital region, as guided by research. The emphasis was on the brain processing visual information and maintaining attention, particularly when the eyes are open and receiving input.

The design was chosen for its suitability in small-sample and exploratory studies, permitting the study of individual changes over time. The four-week intervention period and follow up assessment were chosen to capture both immediate and sustained effects of fractal virtual reality. A randomised waitlist-controlled study is often employed in conjunction with therapeutic interventions. The delayed group provides an untreated comparison for the active group.

ELIGIBILITY:
Inclusion Criteria:

* Must have perceived peri or menopausal symptoms
* Must have normal or corrected to normal hearing and vision
* Must be 18 years or older
* Must have used virtual reality before with no side effects
* Must have a pulse rate of 60 to 80 beats per minute
* Must NOT experience seizures
* Must NOT have coordination difficulties

Exclusion Criteria:

* Do not have peri or menopausal symptoms
* Have coordination difficulties
* Report having claustrophobia
* Pulse rate higher than 80 at rest
* Have sensitivities to flashing lights
* Are prone to migraine
* Have seizures Are younger than 18 years old

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically born women which can include trans men
Enrollment: 18 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Menopause symptoms | 0, 4 and 8 weeks
  This 17 item questionnaire consists of a 4 option (0 not at all, 4 a lot) Likert scale that evaluates menopause symptoms. Example symptoms include difficulty concentrating, loss of interest in sex, pain during sex, and vaginal dryness. Areas are divided into vasomotor symptoms, emotional symptoms, local and sexual symptoms, as well as various physiological symptoms. The Cronbach's alpha is .752. Higher scores indicate higher symptoms of menopause.

SECONDARY OUTCOMES:
Cognitive mindfulness | 0, 4 and 8 weeks
  This is a 10 item questionnaire with 5 response categories (1 never or rarely true through 5 very often always true). Cronbach alpha ranges between 0.69 and 0.76. Subscale scoring is divided into 5 areas, including observing, describing, acting with awareness, non-judging, and non-reactivity. Higher scores reflect higher levels of mindfulness endorsement.
Female Sexual Function Index | 0, 4 and 8 weeks
  This is a 19 item questionnaire on sexual function, including sexual desire, orgasm, lubrication, sexual satisfaction and pain. It has five response categories. Scores include severe 2-7.2, moderate 7.3-14.4, mild to moderate 14.5-21.6, mild 21.7- 28.1 cut-off value, and no female sexual dysfunction 28.2 -36.The lower the score, the higher the level of sexual dysfunction.
The Short Warwick Edinburgh Mental Wellbeing Scale | 0, 4 and 8 weeks
  A 7 item questionnaire with 5 response categories looking at functioning and feeling aspects of wellbeing. The response categories include 1 none of the time to 5 all of the time. There is no reverse scoring. Scores range from 7 to 35 where the latter is the highest level of wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Banbury, Principal Investigator — London Met Uni
Locations (1):
- School of Social Science and Professions, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ma J, Zhao D, Xu N, Yang J. The effectiveness of immersive virtual reality (VR) based mindfulness training on improvement mental-health in adults: A narrative systematic review. Explore (NY). 2023 May-Jun;19(3):310-318. doi: 10.1016/j.explore.2022.08.001. Epub 2022 Aug 5. PMID 36002363
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Result] Feldman, G., Hayes, A., Kumar, S., Greeson, J., & Laurenceau, J. P. (2007). Mindfulness and emotion regulation: The development and initial validation of the Cognitive and Affective Mindfulness ScaleRevised (CAMS-R). Journal of Psychopathology and Behavioral Assessment, 29(3), 177-190
- [Result] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Result] Prause N, Staley C, Roberts V. Frontal alpha asymmetry and sexually motivated states. Psychophysiology. 2014 Mar;51(3):226-35. doi: 10.1111/psyp.12173. Epub 2014 Jan 27. PMID 24460762
- [Result] Ciaurriz Larraz AM, Villena Moya A, Chiclana Actis C. Mindfulness-based intervention and sexuality: a systematic review. Trends Psychiatry Psychother. 2024;46:e20210459. doi: 10.47626/2237-6089-2021-0459. Epub 2023 Feb 20. PMID 36803998
- [Result] Amin SM, El-Gazar HE, Zoromba MA, El-Sayed MM, Awad AGE, Atta MHR. Mindfulness for Menopausal Women: Enhancing Quality of Life and Psychological Well-Being Through a Randomized Controlled Intervention. J Nurs Scholarsh. 2025 Jul;57(4):563-575. doi: 10.1111/jnu.70003. Epub 2025 Feb 24. PMID 39992004
- [Result] Bies AJ, Blanc-Goldhammer DR, Boydston CR, Taylor RP, Sereno ME. Aesthetic Responses to Exact Fractals Driven by Physical Complexity. Front Hum Neurosci. 2016 May 20;10:210. doi: 10.3389/fnhum.2016.00210. eCollection 2016. PMID 27242475